CLINICAL TRIAL: NCT00764790
Title: Immunogenicity and Safety of GSK Biologicals' Thimerosal-free TIV Flu Vaccine Versus a Licensed Comparator in Children
Brief Title: Immunogenicity and Safety of GSK Biologicals' Influenza Vaccine Versus a Licensed Comparator in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111751
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2010-07-27 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluarix; Influenza Vaccines

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (3):
- Fluarix Dose A Group (Experimental): Subjects were administered 1 or 2 doses* of Fluarix vaccine (at Day 0 or at Days 0 and 28) intramuscularly, in the non-dominant upper arm (children >12 months of age) or in the anterolateral thigh (children <12 months of age).
  * Only those subjects who had no history of prior influenza vaccination (i.e. unprimed subjects) received 2 doses.
  Interventions: Biological: Fluarix
- Fluarix Dose B Group (Experimental): Subjects were administered 1 or 2 doses*, half the volume of dose A, of Fluarix vaccine (at Day 0 or at Days 0 and 28) intramuscularly, in the non-dominant upper arm (children >12 months of age) or in the anterolateral thigh (children <12 months of age).
  * Only those subjects who had no history of prior influenza vaccination (i.e. unprimed subjects) received 2 doses.
  Interventions: Biological: Fluarix
- Fluzone Group (Active Comparator): Subjects were administered 1 or 2 doses* of Fluzone vaccine (at Day 0 or at Days 0 and 28) intramuscularly, in the non-dominant upper arm (children >12 months of age) or in the anterolateral thigh (children <12 months of age).
  * Only those subjects who had no history of prior influenza vaccination (i.e. unprimed subjects) received 2 doses.
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluarix — One (Day 0) or two (Day 0 and Day 28) doses by intramuscular injection. Two different doses are tested.
  Arms: Fluarix Dose A Group; Fluarix Dose B Group
Biological: Fluzone — One (Day 0) or two (Day 0 and Day 28) doses by intramuscular injection.
  Arms: Fluzone Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and the safety of GlaxoSmithKline Biologicals' seasonal influenza vaccine, Fluarix, compared to Fluzone (a US-licensed vaccine) in children, 6 to 35 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child aged 6 to 35 months at the time of the first vaccination; children who may or may not have had previous administration of influenza vaccine in a previous season are acceptable.
* Subjects having a parent/guardian who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject's parent/guardian.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the administration of the study vaccine, or planned use during the study period. Routine, registered childhood vaccinations are not an exclusion criterion.
* History of hypersensitivity to any vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* History of Guillain Barré syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* Receipt of an influenza vaccine outside of this study, during current (2008-09) flu season.
* Administration of immunoglobulins and/or blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3317 (Actual)
Dates: Start 2008-10-01; Primary Completion 2009-03-05 (Actual); Study Completion 2009-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (67):
- United States (61):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Conway, Arkansas
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, DeKalb, Illinois
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Cortland, New York
  - GSK Investigational Site, Boone, North Carolina
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Austintown, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Latrobe, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Wexford, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Angelo, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Burke, Virginia
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Li-Kim-Moy J, Wood N, Jones C, Macartney K, Booy R. Impact of Fever and Antipyretic Use on Influenza Vaccine Immune Reponses in Children. Pediatr Infect Dis J. 2018 Oct;37(10):971-975. doi: 10.1097/INF.0000000000001949. PMID 29465480
- [Derived] Pavia-Ruz N, Angel Rodriguez Weber M, Lau YL, Nelson EA, Kerdpanich A, Huang LM, Silas P, Qaqundah P, Blatter M, Jeanfreau R, Lei P, Jain V, El Idrissi M, Feng Y, Innis B, Peeters M, Devaster JM. A randomized controlled study to evaluate the immunogenicity of a trivalent inactivated seasonal influenza vaccine at two dosages in children 6 to 35 months of age. Hum Vaccin Immunother. 2013 Sep;9(9):1978-88. doi: 10.4161/hv.25363. Epub 2013 Jun 19. PMID 23782962
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111751 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111751 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111751 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111751 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111751 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111751 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111751 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Started | 1107 | 1106 | 1104
Completed | 1069 | 1065 | 1074
Not Completed | 38 | 41 | 30
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 10 | 12 | 6
Not completed — Lost to Follow-up | 28 | 29 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group | Total
Number analyzed (Participants) | 1107 | 1106 | 1104 | 3317
Age, Continuous [Mean (Standard Deviation); unit: months] | 20.9 (8.07) | 20.9 (8.42) | 21.0 (8.23) | 20.9 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 539 | 517 | 560 | 1616
  Male | 568 | 589 | 544 | 1701

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Serum Anti-hemagglutinin (HA) Antibodies Against Each of the Influenza Vaccine Strains
Description: GMTs and their 95% confidence interval are presented for all 3 viral strains comprised in the vaccine.
  Post-vaccination timepoints: Day 28 for primed or Day 56 for unprimed subjects
Time Frame: Day 0 (PRE), Day 28 or Day 56 (POST)
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available data.
Measure: Geometric Mean (95% Confidence Interval); unit: titre
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1018 | 1016 | 1031
titre
  A/Brisbane (PRE): number analyzed (Participants) | 1017 | 1013 | 1030
  A/Brisbane (PRE) | 10.4 [9.7 to 11.1] | 10.6 [9.8 to 11.4] | 10.9 [10.1 to 11.7]
  A/Brisbane (POST) | 106.1 [93.8 to 120.1] | 131.6 [116.3 to 148.9] | 232.4 [214.0 to 252.3]
  A/Uruguay (PRE): number analyzed (Participants) | 1017 | 1013 | 1030
  A/Uruguay (PRE) | 12.1 [11.1 to 13.2] | 11.2 [10.2 to 12.2] | 11.6 [10.7 to 12.7]
  A/Uruguay (POST) | 125.6 [113.3 to 139.3] | 158.7 [143.9 to 175.2] | 280.3 [260.3 to 301.9]
  B/Florida (PRE): number analyzed (Participants) | 1017 | 1013 | 1030
  B/Florida (PRE) | 8.4 [7.9 to 9.0] | 8.9 [8.3 to 9.6] | 8.3 [7.7 to 8.8]
  B/Florida (POST) | 113.0 [103.4 to 123.4] | 164.4 [150.2 to 180.1] | 176.4 [162.3 to 191.7]

2. Primary Outcome: Number of Subjects Who Seroconverted
Description: Seroconversion is defined as the number of subjects with either a pre-vaccination anti-HA titer < 1:10 and a post-vaccination titer ≥ 1:40, or a pre-vaccination titer ≥ 1:10 and a minimum 4-fold increase at post-vaccination titer.
  Post-vaccination timepoints: Day 28 for primed or Day 56 for unprimed subjects
Time Frame: Day 28 or Day 56
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1017 | 1013 | 1030
Participants
  A/Brisbane | 636 | 699 | 929
  A/Uruguay | 747 | 808 | 988
  B/Florida | 812 | 864 | 904

3. Secondary Outcome: Number of Seroprotected Subjects
Description: A seroprotected subject is a subject with a serum anti-HA titer
  ≥ 1:40
  Post-vaccination timepoints: Day 28 for primed or Day 56 for unprimed subjects
Time Frame: Day 0 (PRE), Day 28 or Day 56 (POST)
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1018 | 1016 | 1031
Participants
  A/Brisbane (PRE): number analyzed (Participants) | 1017 | 1013 | 1030
  A/Brisbane (PRE) | 185 | 186 | 206
  A/Brisbane (POST) | 699 | 754 | 986
  A/Uruguay (PRE): number analyzed (Participants) | 1017 | 1013 | 1030
  A/Uruguay (PRE) | 222 | 193 | 214
  A/Uruguay (POST) | 788 | 846 | 1012
  B/Florida (PRE): number analyzed (Participants) | 1017 | 1013 | 1030
  B/Florida (PRE) | 171 | 181 | 166
  B/Florida (POST) | 872 | 902 | 935

4. Secondary Outcome: Seroconversion Factor
Description: Seroconversion factor is defined as the fold increase in serum anti-HA GMTs post-vaccination (Day 28 or 56) compared to pre-vaccination (Day 0).
  Post-vaccination timepoints: Day 28 for primed or Day 56 for unprimed subjects
Time Frame: Day 28 or Day 56
Population: Analysis was performed on the ATP cohort for analysis of immunogenicity
Measure: Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1017 | 1013 | 1030
fold increase
  A/Brisbane | 10.2 [9.2 to 11.4] | 12.4 [11.2 to 13.7] | 21.4 [19.9 to 23.1]
  A/Uruguay | 10.4 [9.6 to 11.3] | 14.2 [13.1 to 15.4] | 24.1 [22.6 to 25.7]
  B/Florida | 13.4 [12.4 to 14.5] | 18.4 [17.0 to 20.0] | 21.4 [19.7 to 23.1]

5. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During a 4-day follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, including all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1081 | 1086 | 1090
Participants
  Pain | 403 | 406 | 363
  Redness | 259 | 249 | 253
  Swelling | 152 | 170 | 129

6. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, irritability, loss of appetitie, and temperature.
Time Frame: During a 4-day follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, including all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1080 | 1086 | 1090
Participants
  Drowsiness | 293 | 317 | 298
  Irritability | 386 | 387 | 375
  Loss of appetite | 281 | 273 | 270
  Temperature | 67 | 69 | 72

7. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Time Frame: During a 28-day follow-up period after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1107 | 1106 | 1104
Participants | 565 | 541 | 562

8. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE) and New Onset of Chronic Diseases (NOCD)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
  NOCDs assessed include for example: diabetes, asthma, allergies, autoimmune disease, cancer, neuropathic disorders
Time Frame: During the entire study (Day 0 until Month 6)
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1107 | 1106 | 1104
Participants
  SAE | 35 | 29 | 31
  NOCD | 10 | 8 | 9

9. Secondary Outcome: Number of Subjects Reporting Rare Serious Events
Description: Rare serious events have an occurrence rate of 1/300 (0.3%).
Time Frame: During the entire study (Day 0 until Month 6)
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Number analyzed (Participants) | 1107 | 1106 | 1104
Participants
  Pneumonia | 0 | 0 | 3
  Bronchiolitis | 0 | 3 | 3

ADVERSE EVENTS:
Arm/Group | Fluarix Dose A Group | Fluarix Dose B Group | Fluzone Group
Serious Adverse Events (participants affected / at risk) | 35/1107 | 29/1106 | 31/1104
Other Adverse Events (participants affected / at risk) | 805/1107 | 791/1106 | 808/1104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Dose A Group (N=1107) | Fluarix Dose B Group (N=1106) | Fluzone Group (N=1104)
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 4 | 3 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Croup infectious (Infections and infestations) | 1 | 1 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Electric shock (Injury, poisoning and procedural complications) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 4 | 2
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 2 | 0 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Injury corneal (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 2 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4 | 3
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral rash (Infections and infestations) | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Dose A Group (N=1107) | Fluarix Dose B Group (N=1106) | Fluzone Group (N=1104)
Upper respiratory tract infection (Infections and infestations) | 135 | 116 | 139
Nasopharyngitis (Infections and infestations) | 139 | 119 | 123
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 70 | 60
Pyrexia (General disorders) | 53 | 52 | 62
Diarrhoea (Gastrointestinal disorders) | 62 | 42 | 60
Pharyngitis (Infections and infestations) | 49 | 60 | 52
Pain (General disorders) | 403 | 406 | 363
Redness (General disorders) | 259 | 249 | 253
Swelling (General disorders) | 152 | 170 | 129
Drowsiness (General disorders) | 293 | 317 | 298
Irritability (General disorders) | 386 | 387 | 375
Loss of appetite (General disorders) | 281 | 273 | 270
Temperature (General disorders) | 67 | 69 | 72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.